CLINICAL TRIAL: NCT01554358
Title: Lifestyle and Genetic Factors on Diabetes Risk in Women With GDM After Delivery: Tianjin Gestational Diabetes Prevention Program (TGDPP)
Brief Title: Tianjin Gestational Diabetes Prevention Program (TGDPP)
Acronym: GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Women and Children's Health Center (Other)
Responsible Party: Principal Investigator, HunKun Liu, Project co-investigator, Tianjin Women and Children's Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TWCHC09-01
Record Dates: First submitted 2011-12-13; First posted 2012-03-14 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational diabetes mellitus; Lifestyle intervention
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Other): The women in the intervention group will be given detailed advice about how to achieve the six evidence-based goals of the intervention,7-9 including: 1) reduction in 5-10% of initial body weight in women with body mass index (BMI) ≥24 kg/m2 through the reduction of at least 10% of total calories of their normal meals, 2) total fat intake <30% of energy consumed, 3) carbohydrate intake 55-65% of energy consumed, 4) fiber intake 20-30g per day, and 5) moderate or vigorous exercise for at least 30 min daily, seven days each week.
  Interventions: Behavioral: Lifestyle intervention
- Control (No Intervention): the subjects in the control group had been educated regarding general principles of healthy lifestyle that benefits T2D and obesity prevention, and also informed about the current evidence showing that the lifestyle intervention is effective in women at high risk for T2D during the "run-in" period.

INTERVENTIONS:
Behavioral: Lifestyle intervention — The women in the intervention group will be given detailed advice about how to achieve the six evidence-based goals of the intervention,7-9 including: 1) reduction in 5-10% of initial body weight in women with body mass index (BMI) ≥24 kg/m2 through the reduction of at least 10% of total calories of their normal meals, 2) total fat intake <30% of energy consumed, 3) carbohydrate intake 55-65% of energy consumed, 4) fiber intake 20-30g per day, and 5) moderate or vigorous exercise for at least 30 min daily, seven days each week.
  --------------------------------------------------------------------------------
  Arms: Lifestyle counseling

SUMMARY:
A total of 1,180 women diagnosed with Gestational Diabetes Mellitus (GDM) from 2005 to 2009 and their children have and continues to be randomly assigned to either the intervention group or the control group. A total of 83 women with prior GDM and newly diagnosed diabetes at baseline survey have the nine-month lifestyle intervention program. GDM women in the intervention group will have five consulting sessions with a dietician during the first year and two sessions during the second year. The intervention group are given detailed advice about how to achieve the five goals of the intervention. The primary aim will test whether lifestyle intervention can reduce incident Type 2 Diabetes (T2D) in women with prior GDM. The second aim will test gene-intervention interactions through fine-mapping established genes for glucose, IR, lipids, obesity and T2D in relation to metabolic traits for T2D in GDM women. The third aim will evaluate the effects of the nine-month lifestyle intervention program on cardiovascular risk factors in women with prior GDM and newly diagnosed diabetes. The forth aim will assess if a lifestyle intervention targeting both GDM mothers and their offspring can greatly improve offspring's cardimetablic risk (body weight, glucose and lipid metabolism).

ELIGIBILITY:
Inclusion Criteria for mothers:

1. Age 20-49 years
2. Women diagnosed with GDM between 2005 and 2009.

Inclusion Criteria for children: age 1-5 years at baseline survey.

Exclusion Criteria:

1. Age < 20 and ≥ 50 years
2. Newly diagnosed diabetes in the screening visit
3. The presence of any chronic diseases that could seriously reduce their life expectancy or their ability to participate in the trial
4. Unable or unwilling to give informed consent or communicate with study staff
5. Currently pregnant, or planning to become pregnant in the next four years

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2526 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
incident type 2 diabetes | during 4-year follow-up
Cardiovascular risk factors | 9 month
  Patients with newly diagnosed diabetes in Aim 3
cardimetablic risk | During 4-year follow-up
  Children in Aim 4

SECONDARY OUTCOMES:
approximately 40 SNPs | during 4-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Women's and Children's Health Center, Tianjin, China

REFERENCES:
- [Derived] Li W, Liu H, Feng L, Wang L, Zhang S, Li W, Liu G, Leng J, Shen Y, Gao R, Zhu Y, Yang X, Yu Z, Hu G. Weight change mediates the effect of lifestyle intervention on postpartum diabetes in women with prior gestational diabetes: a secondary analysis of a randomized clinical trial. BMC Med. 2026 Jan 21. doi: 10.1186/s12916-026-04644-y. Online ahead of print. PMID 41559729
- [Derived] Joyce BT, Liu H, Wang L, Wang J, Zheng Y, Nannini D, Drong A, Shiau S, Li W, Leng J, Shen Y, Gao R, Baccarelli A, Hu G, Hou L. Novel epigenetic link between gestational diabetes mellitus and macrosomia. Epigenomics. 2021 Aug;13(15):1221-1230. doi: 10.2217/epi-2021-0096. Epub 2021 Aug 2. PMID 34337972
- [Derived] Liang Z, Wang L, Liu H, Chen Y, Zhou T, Heianza Y, Leng J, Li W, Yang X, Shen Y, Gao R, Hu G, Qi L. Genetic susceptibility, lifestyle intervention and glycemic changes among women with prior gestational diabetes. Clin Nutr. 2020 Jul;39(7):2144-2150. doi: 10.1016/j.clnu.2019.08.032. Epub 2019 Sep 10. PMID 31542245
- [Derived] Chen Y, Liu H, Wang L, Zhou T, Liang Z, Li W, Shang X, Leng J, Shen Y, Hu G, Qi L. Lifestyle intervention modifies the effect of the MC4R genotype on changes in insulin resistance among women with prior gestational diabetes: Tianjin Gestational Diabetes Mellitus Prevention Program. Am J Clin Nutr. 2019 Sep 1;110(3):750-758. doi: 10.1093/ajcn/nqz121. PMID 31271198